CLINICAL TRIAL: NCT03124589
Title: Comparing the Efficacy of an Online Gambling Intervention to a no Intervention Control Condition: Randomized Controlled Trial
Brief Title: Comparing the Efficacy of an Online Gambling Intervention to a no Intervention Control Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 01/19/2017
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Gambling Problem

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): A questionnaire that asks individuals what components of an online intervention they might find useful.
- Online Gambling Internet Intervention (Experimental): An online gambling Internet intervention (housed at CAMH and developed based on the self-help materials created by Professor David Hodgins)
  Interventions: Behavioral: Online Gambling Internet Intervention

INTERVENTIONS:
Behavioral: Online Gambling Internet Intervention — CAMH's online gambling intervention which includes self-help materials as well as a personalized feedback component.
  Arms: Online Gambling Internet Intervention

SUMMARY:
Online interventions for gambling problems hold a strong potential to help people with gambling concerns. However, there are no trials, to-date, that have been able to demonstrate the effectiveness of such an intervention. The current trial will compare participants provided access to an online gambling intervention to those assigned by chance to a no intervention condition in order to test the efficacy of one such Internet intervention for gambling.

Participants will be recruited through Amazon's MTurk crowdsourcing platform. Potential participants identified as problem gamblers who are interested in quitting or reducing their gambling in the next 6 months, or often think about it, based on an initial survey will be invited to complete additional surveys at 6 weeks and 6 months. Those who then agree to be followed up will be randomized to access an online intervention for gambling or a no-intervention website. These participants will then be contacted again at 6 weeks and 6 months to ask about their gambling, and their impressions of the online intervention. The primary hypothesis to be tested is that participants receiving access to the online gambling intervention will report a greater reduction in number of days gambling and in NODS scores at 6-month follow-up than participants in the no intervention control condition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* A score of 5 or over on the Problem Gambling Severity Index (PGSI)
* Thinking about cutting down or quitting their gambling (in next 6 months, or state that they are thinking about it most or almost all of the time)
* Willingness to complete a 6-week and 6-month follow-up survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Change in the variable, National Opinion Research Center DSM Screen for Gambling Problems (NODS) score | Past 6 months
  Screening tool for gambling problems according to DSM-IV criteria

SECONDARY OUTCOMES:
Change in the variable, number of days gambling in the past month | 6 weeks and 6 months
  Total days gambled in the past 30 days
Change in the variable, Gambling Symptom Assessment Scale (GSAS) score | 6 weeks and 6 months
  Gambling symptom severity in the past week

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schell C, Godinho A, Cunningham JA. Examining Change in Self-Reported Gambling Measures Over Time as Related to Socially Desirable Responding Bias. J Gambl Stud. 2021 Sep;37(3):1043-1054. doi: 10.1007/s10899-020-09970-1. PMID 32737814
- [Derived] Cunningham JA, Godinho A, Hodgins DC. Pilot randomized controlled trial of an online intervention for problem gamblers. Addict Behav Rep. 2019 Mar 6;9:100175. doi: 10.1016/j.abrep.2019.100175. eCollection 2019 Jun. PMID 31193792
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research